CLINICAL TRIAL: NCT03982277
Title: A Randomized, Four-arm Open Label Phase Two-b Clinical Trial to Evaluate the Pharmacokinetics, Safety/Tolerability and Efficacy of High Dose Rifampicin in TB-HIV Co-infected Patients on Efavirenz- or Dolutegravir-based Antiretroviral Therapy
Brief Title: Safety and Efficacy of High Dose Rifampicin in Tuberculosis (TB)-HIV Co-infected Patients on Efavirenz- or Dolutegravir-based Antiretroviral Therapy
Acronym: SAEFRIF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST/224/219
Record Dates: First submitted 2019-05-30; First posted 2019-06-11 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-03

CONDITIONS: Tuberculosis
Keywords: High dose rifampicin; TB/HIV co-infected persons; safety; pharmacokinetics; efficacy
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High dose Rifampin + DTG (Experimental): High dose Rifampicin (35mg/kg ) and standard doses of Isoniazid + Ethambutol + Pyrazinamide Dolutegravir based ART regimen
  Interventions: Drug: Rifampin 300 Mg Oral Capsule
- Standard dose Rifampin + DTG (No Intervention): Standard dose rifampicin (10mg/kg) and standard doses of Isoniazid + Ethambutol + Pyrazinamide Dolutegravir based ART regimen
- High dose Rifampin + EFV (Experimental): High dose rifampicin (35mg/kg) and standard doses of Isoniazid + Ethambutol + Pyrazinamide Efavirenz based ART regimen
  Interventions: Drug: Rifampin 300 Mg Oral Capsule
- Standard dose Rifampin + EFV (No Intervention): Standard dose rifampicin (10mg/kg) and standard doses of Isoniazid + Ethambutol + Pyrazinamide Efavirenz based ART regimen

INTERVENTIONS:
Drug: Rifampin 300 Mg Oral Capsule — High dose rifampicin at 35mg/kg
  Arms: High dose Rifampin + DTG; High dose Rifampin + EFV

SUMMARY:
Higher doses of rifampicin has been associated with a faster drop in bacterial load over time, and shorter treatment regimens with high dose rifampicin are being proposed. Sub-therapeutic rifampicin concentrations are common in TB patients and have been demonstrated in several studies carried out among patients with tuberculosis receiving the standard dose (10mg/kg) of rifampicin. Insufficient exposure to isoniazid and rifampicin, which are the cornerstones of TB treatment, has been associated with drug resistance, treatment failure and delayed bacterial clearance from sputum. Evidence has indicated that the current dose of rifampicin (10mg/kg) is inadequate for many patients. Several studies have suggested that dose escalation (to 20-35mg/kg) is safe, and that higher doses (35mg/kg) may accelerate clearance of TB bacteria from the sputum of infected individuals and achievement of target concentrations.15,16 However, these studies have almost entirely been conducted among HIV negative TB patients, or TB-HIV co-infected patients without severe immunosuppression who are not yet receiving antiretroviral therapy (ART). TB-HIV co-infected patients on multiple additional drugs, including ART, are at increased risk of drug-drug interactions and drug related toxicities, including hepatotoxicity. Increasing the dose of rifampicin is a promising approach; however, there is paucity of data on the safety of higher doses of rifampicin in HIV infected patients on ART, and almost no information on the enzyme induction effect of high dose rifampicin on Efavirenz (EFV) and Dolutegravir (DTG). In this study, the investigators will not only evaluate for the enzyme induction effect of 35mg/kg of rifampicin on the most widely used first-line antiretrovirals, but will also look at the safety of these combinations in a population in which there is still scarce safety data. The aim of this study is to determine the safety of higher doses of rifampicin and its effect on the pharmacokinetics of efavirenz and dolutegravir in TB-HIV co-infected patients.

DETAILED DESCRIPTION:
The investigators will enroll 120 TB-HIV co-infected patients initiating TB treatment. Participants will be randomized to either high dose (35mg/kg) or standard dose (10mg/kg) rifampicin in addition to either dolutegravir (DTG) or efavirenz (EFV), for those who are antiretroviral therapy (ART) naïve. Patients who are already on ART will remain on their current ART regimen. The randomization groups (30 participants in each arm) include:Arm One A: R35mg/kg Isoniazid/Ethambutol/Pyrazinamide (HEZ) + DTG, Arm One B: R10mg/kg HEZ + DTG (Control 1), Arm Two A: R35mg/kg HEZ + EFV, Arm Two B: R10mg/kg HEZ + EFV (Control 2).

High dose rifampicin will be administered for the first 8 weeks (intensive phase) of TB treatment. All other anti-TB drugs will be administered at the standard dose using fixed-dose combinations (FDC). All participants will receive standard dose rifampicin during the continuation phase (weeks 9 -24). Pharmacokinetic (PK) blood sampling will be performed after 6 weeks (±2 weeks) of TB treatment. PK sampling will occur pre-dose and at 1, 2, 4 and 8 hours after observed dose for rifampicin and DTG concentrations and approximately 12-14 hours post-dose for EFV (to measure mid-dose interval (MDI) concentration). The EFV MDI and rifampicin pre-dose samples will be collected concurrently in the EFV arms. Safety laboratory tests including liver and renal function tests will be measured every two weeks or when patients present with symptoms suggestive of toxicity. In participants with culture positive TB at baseline, sputum cultures will be performed after 8 weeks of anti-TB treatment.

The investigators will use population pharmacokinetic modelling to determine the rifampicin and DTG exposure in each arm. Using these models the investigators will evaluate for drug-drug interactions between ART and the standard and high dose of rifampicin. Investigators will compare the mid-dose concentrations of EFV and trough concentrations of DTG in each intervention and control arm using Wilcoxon rank-sum test. The investigators will also compare the proportion of participants with grade 3 or 4 adverse events in each arm using the chi-squared test. Investigators will compare the proportion of participants who are sputum culture negative after 8 weeks of treatment among those in the high dose and standard dose arms using the chi-squared test.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Age of ≥18 years
* Confirmed HIV-1 infection
* Already started on EFV-based or DTG-based ART or planned to start on ART
* Diagnosed with tuberculosis and due to initiate rifampicin-containing therapy

Exclusion Criteria:

* Rifampicin resistant TB identified by baseline Xpert Mycobacterium Tuberculous (MTB)/ Rifampicin (RIF)
* Pregnant women or women planning to get pregnant during TB treatment
* Women of reproductive age on DTG who decline the use of effective contraception methods (in particular: intrauterine device or condoms)
* Decompensated liver disease and/or aminotransferases >5x upper limit of normal (ULN)
* Glomerular filtration rate < 50 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Measures of model predicted exposure/pharmacokinetic (PK) parameters | 6 (+/-2) weeks from ART initiation
  Area under the concentration-time curve over 24 hours (AUC(0-24h)) of DTG, EFV and rifampicin, by rifampicin dose (10 vs. 35 mg/kg rifampicin)
Pharmacokinetics of high dose rifampicin on DTG and EFV | 6 (+/-2) weeks from ART initiation
  Maximum concentrations (Cmax), trough concentrations) of DTG, EFV and rifampicin, by rifampicin dose (10 vs. 35 mg/kg rifampicin)

SECONDARY OUTCOMES:
Safety of high dose rifampicin | up to 24 weeks
  Grade 3 or 4 laboratory or clinical adverse events, according to the National Institutes of Health Division of AIDS toxicity tables (DAIDS).
Efficacy of high dose rifampicin | 8 weeks after TB treatment initiation
  Negative sputum cultures

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sekaggya-Wiltshire, MBChB, PhD, Principal Investigator — Infectious Diseases Institute
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) will made available to other researchers for further analysis or met-analysis following direct request to the sponsor (Infectious Diseases Institute).
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication of study results.
Access Criteria: Direct request shall be made to Infectious Diseases Institute for pooling of data and met-analysis

REFERENCES:
- [Background] Milstein M, Lecca L, Peloquin C, Mitchison D, Seung K, Pagano M, Coleman D, Osso E, Coit J, Vargas Vasquez DE, Sanchez Garavito E, Calderon R, Contreras C, Davies G, Mitnick CD. Evaluation of high-dose rifampin in patients with new, smear-positive tuberculosis (HIRIF): study protocol for a randomized controlled trial. BMC Infect Dis. 2016 Aug 27;16(1):453. doi: 10.1186/s12879-016-1790-x. PMID 27567500
- [Background] Diacon AH, Patientia RF, Venter A, van Helden PD, Smith PJ, McIlleron H, Maritz JS, Donald PR. Early bactericidal activity of high-dose rifampin in patients with pulmonary tuberculosis evidenced by positive sputum smears. Antimicrob Agents Chemother. 2007 Aug;51(8):2994-6. doi: 10.1128/AAC.01474-06. Epub 2007 May 21. PMID 17517849
- [Background] Mitchison DA. Role of individual drugs in the chemotherapy of tuberculosis. Int J Tuberc Lung Dis. 2000 Sep;4(9):796-806. PMID 10985648
- [Background] Boeree MJ, Heinrich N, Aarnoutse R, Diacon AH, Dawson R, Rehal S, Kibiki GS, Churchyard G, Sanne I, Ntinginya NE, Minja LT, Hunt RD, Charalambous S, Hanekom M, Semvua HH, Mpagama SG, Manyama C, Mtafya B, Reither K, Wallis RS, Venter A, Narunsky K, Mekota A, Henne S, Colbers A, van Balen GP, Gillespie SH, Phillips PPJ, Hoelscher M; PanACEA consortium. High-dose rifampicin, moxifloxacin, and SQ109 for treating tuberculosis: a multi-arm, multi-stage randomised controlled trial. Lancet Infect Dis. 2017 Jan;17(1):39-49. doi: 10.1016/S1473-3099(16)30274-2. Epub 2016 Oct 26. PMID 28100438
- [Background] Sekaggya-Wiltshire C, von Braun A, Lamorde M, Ledergerber B, Buzibye A, Henning L, Musaazi J, Gutteck U, Denti P, de Kock M, Jetter A, Byakika-Kibwika P, Eberhard N, Matovu J, Joloba M, Muller D, Manabe YC, Kamya MR, Corti N, Kambugu A, Castelnuovo B, Fehr JS. Delayed Sputum Culture Conversion in Tuberculosis-Human Immunodeficiency Virus-Coinfected Patients With Low Isoniazid and Rifampicin Concentrations. Clin Infect Dis. 2018 Aug 16;67(5):708-716. doi: 10.1093/cid/ciy179. PMID 29514175
- [Background] Park JS, Lee JY, Lee YJ, Kim SJ, Cho YJ, Yoon HI, Lee CT, Song J, Lee JH. Serum Levels of Antituberculosis Drugs and Their Effect on Tuberculosis Treatment Outcome. Antimicrob Agents Chemother. 2015 Oct 12;60(1):92-8. doi: 10.1128/AAC.00693-15. Print 2016 Jan. PMID 26459901
- [Background] Burhan E, Ruesen C, Ruslami R, Ginanjar A, Mangunnegoro H, Ascobat P, Donders R, van Crevel R, Aarnoutse R. Isoniazid, rifampin, and pyrazinamide plasma concentrations in relation to treatment response in Indonesian pulmonary tuberculosis patients. Antimicrob Agents Chemother. 2013 Aug;57(8):3614-9. doi: 10.1128/AAC.02468-12. Epub 2013 May 20. PMID 23689725
- [Background] Peloquin CA, Nitta AT, Burman WJ, Brudney KF, Miranda-Massari JR, McGuinness ME, Berning SE, Gerena GT. Low antituberculosis drug concentrations in patients with AIDS. Ann Pharmacother. 1996 Sep;30(9):919-25. doi: 10.1177/106002809603000901. PMID 8876848
- [Background] Sekaggya-Wiltshire C, von Braun A, Scherrer AU, Manabe YC, Buzibye A, Muller D, Ledergerber B, Gutteck U, Corti N, Kambugu A, Byakika-Kibwika P, Lamorde M, Castelnuovo B, Fehr J, Kamya MR. Anti-TB drug concentrations and drug-associated toxicities among TB/HIV-coinfected patients. J Antimicrob Chemother. 2017 Apr 1;72(4):1172-1177. doi: 10.1093/jac/dkw534. PMID 28108678
- [Background] Sloan D. Pharmacokinetic Variability in TB Therapy: Associations with HIV and Effect on Outcome. Paper presented at: Conference on Retroviruses and Opportunistic Infections2014.
- [Background] Chang KC, Leung CC, Yew WW, Kam KM, Yip CW, Ma CH, Tam CM, Leung EC, Law WS, Leung WM. Peak plasma rifampicin level in tuberculosis patients with slow culture conversion. Eur J Clin Microbiol Infect Dis. 2008 Jun;27(6):467-72. doi: 10.1007/s10096-007-0454-6. Epub 2008 Jan 24. PMID 18214560
- [Background] van Ingen J, Aarnoutse RE, Donald PR, Diacon AH, Dawson R, Plemper van Balen G, Gillespie SH, Boeree MJ. Why Do We Use 600 mg of Rifampicin in Tuberculosis Treatment? Clin Infect Dis. 2011 May;52(9):e194-9. doi: 10.1093/cid/cir184. PMID 21467012
- [Background] Boeree MJ, Diacon AH, Dawson R, Narunsky K, du Bois J, Venter A, Phillips PP, Gillespie SH, McHugh TD, Hoelscher M, Heinrich N, Rehal S, van Soolingen D, van Ingen J, Magis-Escurra C, Burger D, Plemper van Balen G, Aarnoutse RE; PanACEA Consortium. A dose-ranging trial to optimize the dose of rifampin in the treatment of tuberculosis. Am J Respir Crit Care Med. 2015 May 1;191(9):1058-65. doi: 10.1164/rccm.201407-1264OC. PMID 25654354
- [Background] Peloquin CA, Velasquez GE, Lecca L, Calderon RI, Coit J, Milstein M, Osso E, Jimenez J, Tintaya K, Sanchez Garavito E, Vargas Vasquez D, Mitnick CD, Davies G. Pharmacokinetic Evidence from the HIRIF Trial To Support Increased Doses of Rifampin for Tuberculosis. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e00038-17. doi: 10.1128/AAC.00038-17. Print 2017 Aug. PMID 28559269
- [Background] Schutz C, Ismail Z, Proxenos CJ, Marais S, Burton R, Kenyon C, Maartens G, Wilkinson RJ, Meintjes G. Burden of antituberculosis and antiretroviral drug-induced liver injury at a secondary hospital in South Africa. S Afr Med J. 2012 Mar 2;102(6):506-11. doi: 10.7196/samj.5650. PMID 22668951
- [Background] Satyaraddi A, Velpandian T, Sharma SK, Vishnubhatla S, Sharma A, Sirohiwal A, Makharia GK, Sinha S, Biswas A, Singh S. Correlation of plasma anti-tuberculosis drug levels with subsequent development of hepatotoxicity. Int J Tuberc Lung Dis. 2014 Feb;18(2):188-95, i-iii. doi: 10.5588/ijtld.13.0128. PMID 24429311
- [Derived] Sekaggya-Wiltshire C, Nabisere R, Musaazi J, Otaalo B, Aber F, Alinaitwe L, Nampala J, Najjemba L, Buzibye A, Omali D, Gausi K, Kengo A, Lamorde M, Aarnoutse R, Denti P, Dooley KE, Sloan DJ. Decreased Dolutegravir and Efavirenz Concentrations With Preserved Virological Suppression in Patients With Tuberculosis and Human Immunodeficiency Virus Receiving High-Dose Rifampicin. Clin Infect Dis. 2023 Feb 8;76(3):e910-e919. doi: 10.1093/cid/ciac585. PMID 35861296
- [Derived] Nabisere R, Musaazi J, Denti P, Aber F, Lamorde M, Dooley KE, Aarnoutse R, Sloan DJ, Sekaggya-Wiltshire C. Pharmacokinetics, SAfety/tolerability, and EFficacy of high-dose RIFampicin in tuberculosis-HIV co-infected patients on efavirenz- or dolutegravir-based antiretroviral therapy: study protocol for an open-label, phase II clinical trial (SAEFRIF). Trials. 2020 Feb 13;21(1):181. doi: 10.1186/s13063-020-4132-7. PMID 32054536
- See also: Published manuscript for results — https://login.research4life.org/tacsgr1academic_oup_com/cid/article/76/3/e910/6647783?login=true